CLINICAL TRIAL: NCT04714333
Title: Detection of COVID-19 by Volatile Organic Compounds in Exhaled Breath (VOCs) - a Pilot Study
Brief Title: Detection of Covid-19 by Volatile Organic Compounds in Exhaled Breath
Acronym: Covid-VOC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Other Study IDs: H20-01234
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our primary aim is to collect breath samples from COVID-19 positive patients at the time of diagnosis, during and after recovery using the same patient as his/her own control to identify VOCs specific to SARS-COV-2 viral infection. A secondary aim is to determine the patient's likely disease trajectory in terms of recovery versus progression to respiratory and or multi-organ failure.

Breath samples will be collected as soon as the patient is admitted to the Vancouver General Hospital COVID Ward with a diagnosis of COVID-19 by RT-PCR in nasopharyngeal/throat swab. A second breath sample will be obtained one week later, or before hospital discharge or if they become sicker prior to transfer to the intensive care. A third sample will be taken to 8-12 weeks after recovery from the illness with a negative COVID-19 RT-PCR test. VOCs in exhaled breath will be measured by gas chromatography-mass spectrometry (GC-TOF-MS or GCxGC-TOFMS). VOC profiles from the symptomatic phase and recovery phase will be compared to determine if there are unique VOCs associated with COVID-19 infection. Comparison of VOC profiles between those who recover and those who progressed will provide information on potential prognostic features. The results of this pilot study will form the basis to determine if a larger study is warranted.

DETAILED DESCRIPTION:
Patients will be recruited from the COVID wards at VGH, all patients admitted will be given a letter of invite on admission if eligible and if interested and eligible will be enrolled. Sample for the study will be collected at the VGH COVID patient wards. Consenting patients and breath collection will be performed in the patients' hospital room with proper personnel protective equipment. A verbal consent will be collected as to not contaminate consent forms. A paper copy will be given or emailed to the participants to have for their own records. .We aim to recruit up to 20 patients. The final number will be dependent on the number of new cases in Vancouver available for the study after REB approval.

Additional participants will be recruited from community testing sites. Participants will be approached to be invited to participate while waiting in their vehicles at the drive-by testing sites.

Breath samples will be analyzed on a SepSolve GC-TOF MS system at the BC Cancer Research Institute.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 18 and 85 years
* Are test positive for COVID-19 (SARS-CoV-2)
* Are capable of providing informed consent to participate in the study

Exclusion Criteria:

* Too sick to provide a breath sample
* Unwilling to sign a consent
* Unwilling to be followed up after you have recovered from the illness.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the COVID wards at VGH, all patients admitted will be given a letter of invite on admission if eligible and if interested and eligible will be enrolled. Consenting patients and breath collection will be performed in the patients' hospital room with proper personnel protective equipment. A verbal consent will be collected as to not contaminate consent forms. We aim to recruit up to 20 patients.
  Additional participants will be recruited from community testing sites. Participants will be approached to be invited to participate while waiting in their vehicles at the drive-by testing sites. If time permits consent and breath collection will be performed while they wait in line. If there is a minimal line up, participant's breath will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-06 (Actual); Primary Completion 2021-05-05 (Estimated); Study Completion 2021-05-05 (Estimated)

PRIMARY OUTCOMES:
Collect breath samples from Covid-19 positive patients at time of diagnosis and post recovery | 6 months
  This is an exploratory trial. The target VOCs are not known at this time. The same patient will be there own control to identify VOCs specific to SARS-CoV-2 viral infection. The presence and absence of VOCs post recovery will indicate the outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Renelle Myers, MD, Principal Investigator — BCCA, Part of the Provincial Health Services Authority
Locations (2):
- Canada (2):
  - BC Cancer Research Centre, Vancouver, British Columbia
  - British Columbia Research Centre, Vancouver, British Columbia